CLINICAL TRIAL: NCT00191867
Title: Assessment of Dose Response of LY333334 in Japanese Postmenopausal Women With Osteoporosis
Brief Title: Clinical Trial of Teriparatide in Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8464; B3D-JE-GHCS
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

INTERVENTIONS:
Drug: Teriparatide

SUMMARY:
The purpose of this study is to assess the Efficacy and Safety of Teriparatide in Japanese Postmenopausal Women with Osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Japanese women with primary osteoporosis
* Postmenopausal women aged at least 55 years
* Patients with a high risk for fracture

Exclusion Criteria:

* History of metabolic bone disorders other than osteoporosis
* History of any secondary causes of osteoporosis
* History of malignant neoplasm within the last 5 years except for superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitively treated
* Severe or chronically disabling conditions other than osteoporosis

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2005-02; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To assess the dose response of LY333334 with the percent change from baseline in lumbar spine mineral density at endpoint

SECONDARY OUTCOMES:
To evaluate the safety of LY333334

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- Japan (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Kagoshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Tokyo

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com